CLINICAL TRIAL: NCT01319916
Title: Open-Label Study to Evaluate the Lipid and Adipokine Profiles Following Subcutaneous Injection of ATX-101 (Sodium Deoxycholate Injection) Into Abdominal Fat Tissue
Brief Title: Lipid and Adipokine Profiles Following Subcutaneous Injection of ATX-101 Into Abdominal Fat Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Daniel R. Lee, M.S., Director, Clinical, Kythera Biopharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-101-10-18
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ATX-101 — ATX-101 2mg/cm2

SUMMARY:
Open Label Study to Evaluate the Serum Lipid and Adipokine Profiles Following Subcutaneous Injection of ATX-101 into Abdominal Fat Tissue

DETAILED DESCRIPTION:
Phase 1, Open Label Study to Evaluate the Serum Lipid and Adipokine Profiles Following Subcutaneous Injection of ATX-101 (Sodium Deoxycholate Injection) into Abdominal Fat Tissue

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy, non-smoking males and nonpregnant, nonlactating females who are 18 to 65 years of age, inclusive, on Day 1A.

  2. Body mass index (BMI) of 18.5 to ≤ 30.0 at within 28 days before the dose of study material.

  3. Stable weight (e.g., approximately ± 10 lbs), in the judgment of the investigator, for at least 3 months before Day 1A.

  4. Sufficient abdominal tissue surface for which 50 injections spaced on 1 cm grid (4 cm x 9 cm square) can be safely administered into fat tissue.

  5. Fasting glucose within normal limits (i.e., 75-100 mg/dL) at within 28 days before the dose of study material.

  6. Fasting hemoglobin A1c within normal limits for the laboratory designated for this trial (e.g., 4 - 5.9%) at within 28 days before the dose of study material.

  7. Fasting triglycerides within normal limits for the laboratory designated for this trial (e.g., < 150m/dL) at within 28 days before the dose of study material.

  8. Fasting cholesterol within normal limits for the laboratory designated for this trial (e.g., < 200 mg/dL) at within 28 days before the dose of study material.

  9. Females must have a negative serum human chorionic gonadotropin (hCG) test result from a sample obtained within 28 days before the beginning of the confinement period and again after admission to the research facility for the confinement period, but before the dose of study material. Females must agree to practice adequate contraception, in the judgment of the investigator, during the course of the trial.

  10. Negative hepatitis B, hepatitis C, and HIV test results. 11. The subject is expected to comply with and understand the visit schedule and all of the protocol-specified tests and procedures.

  12. The subject is medically able to undergo the administration of study material as determined by clinical and laboratory evaluations obtained within 28 days before Day 1A for which the investigator identifies no clinically significant abnormality.

  13. Signed informed consent obtained before any study-specific procedure is conducted

Exclusion Criteria:

* 1. History of any intervention (e.g., liposuction) or trauma associated with the abdominal area, which in the judgment of the investigator, may affect subject's safety or other evaluations of treatment.

  2. Subjects who, for any reason, are on active diet, calorie restriction, or attempting to lose weight.

  3. Blood donation of 500 mL or blood transfusion within 60 days before Day 1A, or plasma donation within 7 days before Day 1A.

  4. Diagnosis of lipodosis (e.g., Gaucher, Niemann-Pick, or Fabry disease) or other confounding metabolic diseases.

  5. History of hypertriglyceridemia (triglycerides > 200 mg/dL), hypercholesterolemia (cholesterol > 240 mg/dL), or hyperlipidemia.

  6. Use of statins (e.g., Vitorin, Lipitor, Lopid) or other lipid-lowering agent (e.g., nicotinic acid) within 28 days or five (5) half-lives, whichever is greater, before Day 1A.

  7. History of diabetes or screening results indicative of diabetes. 8. Use of antiglycemic agents at any time before screening. 9. Use of any medication that results in systemic exposure beginning during the screening period.

  10. Any medical condition (e.g., respiratory, cardiovascular, renal, hepatic, neurological disease, uncontrolled hypertension, thyroid dysfunction) that would interfere with laboratory or safety assessments, compromise the ability of the subject to undergo study procedures, or compromise the subject's ability to give informed consent.

  11. Treatment with oral anticoagulants (e.g., warfarin, heparin) within 10 days before Day 1A; anticipated need for agents with anticoagulative effects during the course of the trial.

  12. History of sensitivity to any components of the study material or topical anesthetics (e.g., lidocaine, benzocaine, novocaine).

  13. Previous enrollment into this trial or treatment with ATX-101 or agents containing deoxycholate.

  14. Treatment with an investigational agent within 28 days before Day 1A.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Effects of ATX-101 on serum lipid and deoxycholate
  acute effects of ATX-101 on serum lipid and deoxycholate profile following subcutaneous administration into abdominal fat tissue.

SECONDARY OUTCOMES:
Adipokine levels following subcutaneous administration of ATX-101
  To evaluate adipokine levels following subcutaneous administration of ATX-101 into abdominal fat tissue

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD, PhD, Study Director — Kythera Biopharmaceuticals
Locations (1):
- Robert Cooper, M.D. Cetero Research, Fargo, North Dakota, United States